CLINICAL TRIAL: NCT06451432
Title: 'Hernia Endoscopic oR opeN Repair In chIldren Analysis": A Randomized Controlled Trial to Study the (Cost-) Effectiveness of Paediatric Laparoscopic Hernia Repair Compared to Open Hernia Repair
Brief Title: The (Cost-) Effectiveness of Paediatric Laparoscopic Hernia Repair Compared to Open Hernia Repair
Acronym: HERNIIA-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Sanne Maat, Coördinating investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL71765.029.20
Record Dates: First submitted 2024-05-27; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Inguinal Hernia
Keywords: pediatric; PIRS; open inguinal hernia repair
MeSH Terms: conditions — Hernia, Inguinal | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing two study groups
Masking Description: Due to the nature of the intervention (different type of scars), masking is not possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Percutaneous Inguinal Ring Suturing (PIRS) technique
  Interventions: Procedure: Percutaneous Inguinal Ring Suturing (PIRS) technique
- Control group (No Intervention): Open inguinal hernia repair

INTERVENTIONS:
Procedure: Percutaneous Inguinal Ring Suturing (PIRS) technique — Percutaneous Inguinal Ring Suturing (PIRS) technique
  Arms: Intervention group

SUMMARY:
This study assess the (cost-)effectiveness of open versus laparoscopic Percutaneous Inguinal Ring Suturing (PIRS) technique for unilateral inguinal hernia repair in children aged 0-16 years.

DETAILED DESCRIPTION:
Research question Inguinal hernia repair is one of the most common operations in children. After open unilateral inguinal hernia repair, 6-8% of patients develops an inguinal hernia on the contralateral side. Laparoscopic inguinal hernia offers the opportunity to inspect the contralateral groin and repair an asymptomatic contralateral hernia, if present.

Main question: What is the most (cost-)effective treatment strategy for unilateral inguinal hernia repair in children aged 0-16 years: the open or laparoscopic Percutaneous Inguinal Ring Suturing (PIRS) technique?

Hypothesis The optimal treatment for children with an inguinal hernia is laparoscopic hernia repair, since the surgeon can inspect and possibly, repair, the contralateral groin. Laparoscopic inguinal hernia repair results in less operations and exposure to anaesthesia, less hospital admissions, lower costs and a better quality of life compared to open inguinal hernia repair.

Study design Multicentre randomized controlled trial.

Study population Children aged 0 - 16 years with a unilateral inguinal hernia.

Intervention Inguinal hernia repair with the laparoscopic PIRS technique.

Usual care/comparison Inguinal hernia repair with the open technique.

Outcome Measures Primary: Number of operations related to inguinal hernia repair and cost-effectiveness (social and healthcare related costs). Secondary: complications, total duration of surgery (including anaesthesia and total duration of operating room time), post-operative pain, length of hospital stay, time to normal daily activities, cosmetic appearance, health-related quality of life. All outcome measures will be assessed within two years after the primary inguinal hernia correction.

Sample size/data analysis 464 patients (power of 0.80, alpha 0.05). Cost-effectiveness analysis/budget impact analysis The economic evaluation will be assessed from a societal and health care perspective. Cost-effectiveness will be assessed in terms of QALYs and the primary and secondary outcomes. A budget impact analysis will be conducted using the "Budget Impact Analyse - leidraad en rekentool" of ZonMw. Missing data will be imputed.

ELIGIBILITY:
Inclusion Criteria:

1. Infants aged 0 months to 16 years of age with a primary unilateral inguinal hernia undergoing hernia repair

Exclusion Criteria:

1. incarcerated inguinal hernia, which have to be operated immediately,
2. recurrent hernia
3. ventricular-peritoneal drain
4. non-descended testis
5. parents who are not able to understand the nature or consequences of the study.

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 464 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Re-operation rate | within two years after the primary inguinal hernia repair
  Number of re-operations related to primary inguinal hernia repair

SECONDARY OUTCOMES:
Complications | Within two years after the primary inguinal hernia repair
  Surgical and anesthesiological complications
Duration of Surgery | Within two years after the primary inguinal hernia repair
  Total duration of surgery (including anaesthesia and total duration of operating room time)
Post-operative pain | Within two years after the primary inguinal hernia repair
  Postoperative pain is as medication requirement and VAS-score (1-9 score, 9 point scale, higher score equals more pain)
Length of hospital stay | Within two years after the primary inguinal hernia repair
  Number of days
Time to normal daily activities | Within two years after the primary inguinal hernia repair
  Number of days
Cosmetic appearance | Within two years after the primary inguinal hernia repair
  Cosmetic appearance is scored by parents and a member of a research team using a 5-Likert scale (scale 1-5, higher score equals a better outcome)
Health-related quality of life | Within two years after the primary inguinal hernia repair
  Health related quality of life will be measured using the EQ-5D version (EQ-5D-5L) four weeks, one year, and two years after primary surgery. A higher score equals a better outcome.
Cost-effectiveness | Cost-effectiveness is measured qithin two years after the primary inguinal hernia repair
  Cost-effectiveness is based of societal and healthcare costs.

CONTACTS AND LOCATIONS:
Overall Officials: Joep Derikx, prof.dr., Principal Investigator — Amsterdam UMC
Locations (9):
- Netherlands (9):
  - Maxima Medisch Centrum, Veldhoven, North Brabant
  - FlevoZiekenhuis, Almere, North Holland
  - Amsterdam UMC, locatie AMC and VUmc, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland
  - MST, Enschede, Twente
  - Alrijne Ziekenhuis, Leiderdorp, Zuid-hHolland
  - UMCG, Groningen
  - Maastricht UMC+, Maastricht
  - Isala Ziekenhuis, Zwolle

REFERENCES:
- [Derived] Maat SC, de Vreeze LE, Eurlings R, Anema J, Van Baren R, Been JV, van den Broek F, Cakir H, van Dongen JM, Ferenschild F, de Graaf J, Nijveldt R, Ottenhof A, Ploeg AJ, Rippen H, Ruiterkamp J, Twisk JWR, Vermeulen E, De Wit R, Zijp G, van Heurn ELW, Derikx JPM. HERNIIA-II trial (Hernia Endoscopic oR opeN repair In chIldren Analysis): a protocol of a multicentre randomised controlled trial to study the (cost-)effectiveness of laparoscopic hernia repair compared to open hernia repair in children 0-16 years. BMJ Open. 2025 Dec 4;15(12):e110662. doi: 10.1136/bmjopen-2025-110662. PMID 41344705